CLINICAL TRIAL: NCT01269437
Title: Open-label, Randomized, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Budesonide Novolizer Dry Powder Inhaler Compared With Budesonide Turbuhaler Dry Powder Inhaler in Chinese Mild to Moderate Asthma Patients
Brief Title: Efficacy and Safety Study of Budesonide Novolizer Dry Powder Inhaler 200μg to Treat Chinese Patients With Mild to Moderate Asthma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NovaMed Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM2010002
Record Dates: First submitted 2010-12-31; First posted 2011-01-04 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-04

CONDITIONS: Asthma
Keywords: mild to moderate asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide, Novolizer (Experimental): Budesonide Dry Powder Inhaler
  Interventions: Drug: Budesonide dry powder inhaler
- BudesonideTurbuhaler (Active Comparator): Budesonide Dry Powder Inhaler
  Interventions: Drug: Budesonide dry powder inhaler

INTERVENTIONS:
Drug: Budesonide dry powder inhaler — 200mcg per inhalation, twice daily, for 12 weeks

SUMMARY:
This is an open-label, randomized, parallel Group, multicenter study to evaluate the efficacy and safety of budesonide novolizer dry powder inhaler compared with budesonide turbuhaler dry powder inhaler in Chinese mild to moderate asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent by the subject and his/her legal guardian if the subject is under 18 years old.
* Male or females aged more than 12 and under 70
* Had a definite diagnosis of asthma with symptoms of cough/expectoration/chest tightness/wheeze/breathlessness within the last one month
* Inhaled corticosteroid (ICS) naïve or no regular use of ICS within the last one month (It is suggested that ICS average daily dose with no more than 100mg budesonide or equal within the last month as "No-regular-use")
* FEV1 between 60% and 85% of predicted normal values
* Reversibility test of airway obstruction is positive, i.e. degree of reversibility in FEV1 as over 12%(included) and 200ml(included). Or average diurnal PEFR variability is not less than 20% in two weeks.
* Are able to use Peak Flow Meter and record it on patient diary card

Exclusion Criteria:

* Asthma exacerbation leading to hospitalization for more than 2 days within the last 6 months or emergency room visit due to asthma exacerbation in the last 3 months prior to screening
* Infection of respiratory system in the last 4 weeks prior to screening visit
* Use of oral, injectable, rectal or transdermal glucocorticoid in the last 4 weeks prior to screening visit
* Use of Leukotriene receptor antagonist (LTRAs), oral b2 agonist, methylxanthines or use of inhaled long acting b2 agonist, inhaled anticholinergic receptor in the last 1 week, or inhaled Tiotropium Bromide within 45 days prior to screening visit
* Patients with chronic obstructive pulmonary disease (COPD)or COPD with asthma
* Patients with severe persistent asthma (Based on definition in GINA 2006)
* Patients with specific immunity treatment (including monoclonal antibody treatment) due to asthma within the 6 months prior to screening visit
* Patients with eye disorders including cataract, glaucoma and herpes virus infection
* Smoking history of 10 pack-year (1 pack-year refers to 20 cigarette per day for 1 year)
* History of drug or alcohol abuse
* History of adrenal disease
* History of malignancy disease in the last 5 years, with the exception of basal cell carcinoma
* Heart function failure or any severe systematic disease, at the investigator's discretion, which will make it undesirable for the patient to participate in the trial or which could jeopardize compliance with the trial protocol
* ALT or AST > 2 times of upper limit of reference range
* Creatinine (Cr) > 159µmol/L for males or > 141µmol/L for females
* Patients with hypersensitivity to budesonide and/or lactose
* Participation in a clinical study or treatment with a non-approved experimental medication in the last 1 month
* Pregnant or breast-feeding women, or women of childbearing age without appropriate contraception measures

Limitations:

The following medications are prohibited from screening onward:

* Use of oral, injectable, rectal or transdermal glucocorticoid
* Inhaled nedocromil sodium/Inhaled cromoglycate sodium
* Leukotriene receptor antagonist
* Methylxanthines
* Inhaled long acting b2 agonist
* Oral b2 agonist
* Inhaled anticholinergic receptor
* Any b2 receptor blocker (Including eye drops)

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of budesonide delivered by Novolizer to that delivered by Turbuhaler in terms of mPEF （morning peak expiratory flow） in Chinese mild to moderate asthma patients | 12 weeks
  The change of mPEF in the Week 11-12 of treatment from baseline

SECONDARY OUTCOMES:
To evaluate the improvement of FEV1(Forced Expiratory Volume in One Second) in Chinese mild to moderate asthma patients after treatment of budesonide delivered by Novolizer or Turbuhaler | 12 weeks
  The change of FEV1 in the Week 12 of treatment from baseline
To evaluate the improvement of ePEF （Evening Peak Expiratory Flow） in Chinese mild to moderate asthma patients after treatment of budesonide delivered by Novolizer or Turbuhaler | 12 weeks
  The change of ePEF in the Week 11-12 of treatment from baseline
To evaluate the improvement in ACT (Asthma Control Test) score in Chinese mild to moderate asthma patients after treatment of budesonide delivered by Novolizer or Turbuhaler | 12 weeks
  The change of ACT scores in the Week 12 of treatment from baseline
To evaluate the tolerability and safety of budesonide delivered by Novolizer or Turbuhaler in Chinese mild to moderate asthma patients | 15 weeks
  It will be assessed according to numbers of adverse event and laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue BAI, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (11):
- China (11):
  - The Second Artillery General Hospital of PLA, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Foshan, Foshan, Guangdong
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong
  - Zhongda Hospital of Southeast University, Nanjing, Jiangsu
  - Shengjing Hospital, Shenyang, Liaoning
  - Dongfang Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Putuo District Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The General Hospital of Shenyang Military Region, Shenyang, Shenyang